CLINICAL TRIAL: NCT02496507
Title: A Mixed-methods Evaluation of Sit-stand Workstations in an Office Setting: a Randomised Controlled Trial
Brief Title: A Mixed-methods Evaluation of Sit-stand Workstations in an Office Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Lee Graves, Lecturer/Senior Lecturer, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-SPS-Graves1
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Physical Activity
Keywords: sitting; intervention; desks; workplace; cardiovascular; metabolic; qualitative; randomised controlled trial
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Provision of a sit-stand workstation for use at work.
  Interventions: Other: Sit-stand workstation
- Control (No Intervention): Participants were asked to maintain their normal work practices and received no intervention. Participants were offered the opportunity to have a sit-stand workstation installed for 8 weeks after all data collection.

INTERVENTIONS:
Other: Sit-stand workstation — After baseline, each participant had a sit-stand workstation installed on their existing workplace desk. A single or dual monitor WorkFit-A with Worksurface+ workstation was installed, dependent on the number of monitors. The monitor(s) and keyboard were housed on the workstation and the workstation could be quickly raised up and down by hand to enable seated or standing work. Participants were not prescribed an amount of time to use the station. Ergotron Ltd provided and installed the workstations and gave participants basic face-to-face training and ergonomic information on correct use. Participants received a web link to manufacturer ergonomic guidelines via an email from the research team. After end-intervention data collection, manufacturer staff uninstalled the workstations.
  Arms: Intervention

SUMMARY:
The purpose of this study is to investigate whether a device that allows office workers to sit or stand whilst working can reduce their sitting time at work and improve their health over 8 weeks.

DETAILED DESCRIPTION:
Study design

Treatment arms in this two-arm parallel-group randomised controlled trial (RCT) included a sit-stand workstation intervention group (each participant received a sit-stand workstation) and a control group (usual practice).

Recruitment

- Organisation level

Office workers from one organisation were targeted by the research team in August-September 2013. Consent was sought from 11 departmental managers for employee recruitment, installation of sit-stand workstations, study contact and laboratory visits during work time. Departments were located across four buildings with varying office layout (open-plan, individual offices or a combination). Employees within the targeted departments were predominantly administrative staff.

- Individual level

Via an email from the research team, all employees in consenting departments received an overview of the study and participant information sheet, and were invited to a study information session (two sessions were organised per department). Employees were given 2 weeks to express interest. Interested employees were screened for eligibility using stated criteria by the research team via telephone. If inclusion criteria were met, written informed consent was obtained and baseline assessments scheduled. There was no racial or gender bias in the selection of participants.

Group assignment and Intervention

Following baseline assessments, participants were assigned by one member of the research team to a treatment arm using a randomised block design and random number table. Departments served as blocks and participants within departments were randomly assigned at the individual-level to an arm. Assignment of individual participants within each department alternated between arms (i.e. intervention, control, intervention, control…).

Data collection

At baseline, 4 weeks (mid-intervention) and 8 weeks (end-intervention), participants' office-based behaviours were assessed via ecological momentary assessment (EMA) diaries. At baseline and 8 weeks, participants attended University laboratories in the morning for individual assessments of other stated outcomes. Prior to laboratory visits, participants were required to fast for a minimum of 8 hours, avoid the consumption of alcohol for 12 hours, and avoid strenuous exercise for 24 hours.

Sample size

Allowing for small drop out, the study aimed to recruit 25 participants per arm, and retain 23 participants per arm. A sample size of 23 per arm was chosen a priori to achieve 90% power (alpha 5%; two-tailed) to detect a minimum difference of 60 minutes/8-hour workday between arms for workplace sitting time (primary outcome: expected SD of 60 minutes/day). Data collection for vascular and metabolic outcomes would provide effect size estimates for power calculations in subsequent trials.

Statistical analyses

* Data was analysed using the Statistical Package for the Social Sciences (SPSS) version 22 (IBM, New York, USA) with the alpha level set at p≤0.05. Intervention effects were compared at 4 weeks (sitting, standing and walking) and 8 weeks (all outcomes) from baseline using analysis of covariance (ANCOVA). The variable change score (4 or 8 weeks minus baseline) was the dependent variable, with intervention arm (control vs intervention) the independent variable. In all analyses, covariates were the baseline value for the variable to control for any imbalances at baseline. Anthropometric, sociodemographic, work-related and office-environment characteristics were tested as potential confounders for all outcomes. Confounders were entered as covariates if significant associations (p≤0.05) were observed with changes in an outcome and the effect on the mean difference between groups exceeded 20%. For changes in sitting, standing and walking time, baseline values of the other two behaviours were tested as potential confounders, though no effects on the mean difference between groups exceeded 20%. Adjusted change scores and 95% confidence intervals (CIs) for the difference in change between groups are presented unless stated otherwise. Acceptability and feasibility data are reported as medians and quartiles.
* Missing data and Intention-to-treat analysis Due to participant withdrawal, lost EMA diaries or the inability to conduct assessments, data were missing for all outcomes. Accordingly, a per-protocol analysis was conducted and participants were excluded from analyses for outcomes they were missing data for. For workplace sitting, standing and walking, the per-protocol analysis was compared with an intention-to-treat analysis, as a sensitivity analysis. To treat missing data, the fully conditional imputation technique and ten imputation sets were used due to a low rate of missing data. Imputation was based on all 47 randomized participants.
* Minimum important differences analysis Inferential statistics were ran using minimum clinically important difference principles, described elsewhere. Briefly, this approach makes inferences based on meaningful magnitudes and is recommended alongside hypothesis testing. A spreadsheet computed the quantitative and qualitative probability that the true effects were beneficial, trivial or harmful, after the outcome statistic, its p value, and the smallest/minimal important difference was entered. Minimum important differences for sitting and standing were 60 minutes/day, and for walking 10 minutes/day. Minimum important differences for other outcomes were determined through a distribution-based method as a Cohen's d (standardized difference between change scores between groups) of 0.2 between-subjects standard deviations (SDs). The SD of pooled baseline data was used to negate the possibility of individual differences from the intervention influencing the SD at 8 weeks. For each effect at 8 weeks, quantitative probabilities for benefit, trivial and harm, and qualitative descriptors are reported. Effects were interpreted as unclear if probabilities for benefit and harm were >5%.

ELIGIBILITY:
Inclusion Criteria:

* full-time member of staff
* access to a work telephone and desktop computer with internet

Exclusion Criteria:

* have a cardiovascular or metabolic disease
* taking any medication
* pregnant
* planned absence > 1 week during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in workplace sitting time at 4 and 8 weeks | Baseline (week 0), Mid-intervention (4 weeks), End-intervention (8 weeks)
  An ecological momentary assessment (EMA) diary assessed time spent sitting, standing, walking and in other activities during work hours over 5 days (Monday-Friday). At 15-minute intervals participants used a diary to record their main behaviour in response to the question: "What are you doing right now?" The options were sitting, standing, walking or other. If other was selected, participants were instructed to write the activity they were doing.
  Time spent in each behaviour per day was estimated by multiplying the frequency of recordings by 15. A diary day was considered valid if data entries were provided for ≥75% of time spent at work. Time spent in each behaviour was calculated for each valid day and means were calculated from valid days. To be retained for analyses, participants had to provide ≥2 valid days at each time point.

SECONDARY OUTCOMES:
Change from baseline in workplace standing time at 4 and 8 weeks | Baseline (week 0), Mid-intervention (4 weeks), End-intervention (8 weeks)
  An ecological momentary assessment (EMA) diary assessed time spent sitting, standing, walking and in other activities during work hours over 5 days (Monday-Friday). At 15-minute intervals participants used a diary to record their main behaviour in response to the question: "What are you doing right now?" The options were sitting, standing, walking or other. If other was selected, participants were instructed to write the activity they were doing.
  Time spent in each behaviour per day was estimated by multiplying the frequency of recordings by 15. A diary day was considered valid if data entries were provided for ≥75% of time spent at work. Time spent in each behaviour was calculated for each valid day and means were calculated from valid days. To be retained for analyses, participants had to provide ≥2 valid days at each time point.
Change from baseline in workplace walking time at 4 and 8 weeks | Baseline (week 0), Mid-intervention (4 weeks), End-intervention (8 weeks)
  An ecological momentary assessment (EMA) diary assessed time spent sitting, standing, walking and in other activities during work hours over 5 days (Monday-Friday). At 15-minute intervals participants used a diary to record their main behaviour in response to the question: "What are you doing right now?" The options were sitting, standing, walking or other. If other was selected, participants were instructed to write the activity they were doing.
  Time spent in each behaviour per day was estimated by multiplying the frequency of recordings by 15. A diary day was considered valid if data entries were provided for ≥75% of time spent at work. Time spent in each behaviour was calculated for each valid day and means were calculated from valid days. To be retained for analyses, participants had to provide ≥2 valid days at each time point.
Change from baseline in flow-mediated dilation (FMD) at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  A measure of endothelial dysfunction, which is an early and integral manifestation of atherosclerotic disease.
Change from baseline in carotid artery intima media thickness (cIMT) at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  An early subclinical marker of structural atherosclerosis.
Change from baseline in plasma glucose at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Assessed via standard venepuncture technique
Change from baseline in triglycerides at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Assessed via standard venepuncture technique
Change from baseline in total cholesterol at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Assessed via standard venepuncture technique
Change from baseline in musculoskeletal discomfort or pain at the neck/shoulders at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Assessed via an adapted questionnaire from a previous trial
Change from baseline in musculoskeletal discomfort or pain at the lower back at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Assessed via an adapted questionnaire from a previous trial
Change from baseline in musculoskeletal discomfort or pain at the upper back at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Assessed via an adapted questionnaire from a previous trial
Change from baseline in body mass index at 8 weeks | Baseline (week 0), End-intervention (8 weeks)
  Calculated from assessment of stature and body mass
Acceptability of the sit-stand workstation | End-intervention (8 weeks)
  (Intervention arm only) Assessed via a 19-item five-point Likert scale (1 strongly disagree, 2 disagree, 3 neutral, 4 agree, 5 strongly disagree) adapted from a previous trial.
Feasibility of the sit-stand workstation | End-intervention (8 weeks)
  (Intervention arm only) Assessed via a 19-item five-point Likert scale (1 strongly disagree, 2 disagree, 3 neutral, 4 agree, 5 strongly disagree) adapted from a previous trial.
Acceptability of the sit-stand workstation | End-intervention (8 weeks)
  (Intervention arm only) Interviews
Feasibility of the sit-stand workstation | End-intervention (8 weeks)
  (Intervention arm only) Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Lee EF Graves, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Result] Batterham AM, Hopkins WG. Making meaningful inferences about magnitudes. Int J Sports Physiol Perform. 2006 Mar;1(1):50-7. PMID 19114737
- [Result] Hopkins WG, Marshall SW, Batterham AM, Hanin J. Progressive statistics for studies in sports medicine and exercise science. Med Sci Sports Exerc. 2009 Jan;41(1):3-13. doi: 10.1249/MSS.0b013e31818cb278. PMID 19092709
- [Derived] E F Graves L, C Murphy R, Shepherd SO, Cabot J, Hopkins ND. Evaluation of sit-stand workstations in an office setting: a randomised controlled trial. BMC Public Health. 2015 Nov 19;15:1145. doi: 10.1186/s12889-015-2469-8. PMID 26584856